CLINICAL TRIAL: NCT04005495
Title: Emory Teaching Kitchen Collaborative
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Ardmore Institute of Health (Other)
Responsible Party: Principal Investigator, Sharon Horesh Bergquist, Assistant Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB00109546
Record Dates: First submitted 2019-06-27; First posted 2019-07-02 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Healthy Lifestyle
Keywords: Kitchen Collaborative; Healthful habits; Worksite wellness program; Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Teaching kitchen program (Experimental): The teaching kitchen model is an innovative, multidisciplinary approach for motivating and establishing healthful habits and behaviors. The program combines didactic information with experiential learning in nutrition, culinary arts, exercise, yoga, and mindfulness.
  Interventions: Behavioral: Teaching kitchen program

INTERVENTIONS:
Behavioral: Teaching kitchen program — The teaching kitchen program will include five 4-hour Saturday classes every other weekend over the course of 10 weeks (5 sessions totaling 20 hours of instruction). It will be taught by subject matter experts from the Emory University faculty and staff as well as potentially from the community. The classes will include the scientific rationale, practical applications, and recommendations for implementing self-care components into participants' daily lives. Experiential learning will include hands-on cooking demonstrations, mindfulness-based lunches, a yoga session, and a group exercise session. Rather than being prescriptive, the lectures and demonstrations are geared to inspire self-designed and personalized alterations in dietary patterns and behaviors that will match participants' culture, preferences, and health conditions. Biometrics and survey instruments will be assessed at 4 times: at baseline, after the 10-week program, and at 6 and 12 months after the program.

SUMMARY:
The aim of the project is to evaluate the feasibility and acceptance of a teaching kitchen program as a worksite wellness program at Emory University

DETAILED DESCRIPTION:
The teaching kitchen model is an innovative, multidisciplinary approach for motivating and establishing healthful habits and behaviors. The self-care program combines didactic information with experiential learning in nutrition, culinary arts, exercise, yoga, and mindfulness. The aim of the project is to evaluate the feasibility and acceptance of teaching kitchen program as a worksite wellness program at Emory University. Changes in biomarkers and self-reported behaviors will be evaluated up to one year.

ELIGIBILITY:
Inclusion Criteria:

* age 18-65
* body mass index greater than or equal to 30,
* willingness to appear in videotapes and photographs that will be obtained during the course of the teaching kitchen program
* preference will be given to those with a cardiometabolic risk factor, such as diabetes mellitus, hypertension, and/or hyperlipidemia.

Exclusion Criteria:

* any health condition that would limit participation, including bariatric surgery, pregnancy, cardiovascular, pulmonary, orthopedic or neurologic medical problem, or gluten or nut allergy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2019-07-17 (Actual); Primary Completion 2021-05-04 (Actual); Study Completion 2021-05-04 (Actual)

PRIMARY OUTCOMES:
Percent of enrolled participants attending 2-week visit | 2-week visit
  Program attendance will be assessed by calculating percent of enrolled participants completing the program visits
Percent of enrolled participants attending 4-week visit | 4-week visit
  Program attendance will be assessed by calculating percent of enrolled participants completing the program visits
Percent of enrolled participants attending 6-week visit | 6-week visits
  Program attendance will be assessed by calculating percent of enrolled participants completing the program visits
Percent of enrolled participants attending 8-week visit | 8-week visit
  Program attendance will be assessed by calculating percent of enrolled participants completing the program visits
Percent of participants completing the program | 10-week visit
  Program completion will be assessed by calculating percent of participants completing the program

SECONDARY OUTCOMES:
Change in RAND Health 36-Item scale score | Baseline, 10-week, and 6 and 12 months after the program
  RAND Health 36-Item scale is used to evaluate global health, quality of life, and presenteeism. All items are scored so that a high score defines a more favorable health state. In addition, each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively. Scores represent the percentage of total possible score achieved.
Change in frequency of absence from work | Baseline, 10-week, and 6 and 12 months after the program
  A single question will be asked about the frequency of absence from work
Change in percent body fat | Baseline, 10-week, and 6 and 12 months after the program
  Body composition will be measured by seca medical Body Composition Analyzer (mBCA) 515. This device utilizes 8-point Bioelectrical Impedance Analysis to assess percent body fat. This is a non-invasive technique, taking about two minutes, that requires standing on a scale.
Change in BMI | Baseline, 10-week, and 6 and 12 months after the program
  Body Mass Index (BMI) is a person's weight in kilograms divided by the square of height in meters.
Change in systolic blood pressure | Baseline, 10-week, and 6 and 12 months after the program
  Blood pressure will be measured using blood pressure monitor
Change in diastolic blood pressure | Baseline, 10-week, and 6 and 12 months after the program
  Blood pressure will be measured using blood pressure monitor
Change in Dietary Intake score | Baseline, 10-week, and 6 and 12 months after the program
  Dietary Intake will be assessed using the 8-item Starting The Conversation brief dietary assessment and intervention tool for health professionals. Response options for the survey items are organized into three columns: the left column indicates the most healthful dietary practices (scored 0); the center column indicates less healthful practices (scored 1); and the right column indicates the least healthful practices (scored 2). Item scores are added to create a summary score (range 0-16), with lower summary scores reflecting a more healthful diet and higher scores reflecting the greatest room for improvement.
Change in Cooking Habits score | Baseline, 10-week, and 6 and 12 months after the program
  Cooking Frequency and Confidence questionnaire - items 1,2, 8- will be used to assess change in habits pre to post intervention.Responses range on a scale of 1-6. Higher score reflects more favorable state and lower score reflects the greatest room for improvement.
Change in Cooking Confidence score | Baseline, 10-week, and 6 and 12 months after the program
  Cooking Frequency and Confidence questionnaire will be used to assess confidence to prepare new recipes from basic ingredients. Items 3-7 (assessing cooking confidence) are scored on a scale of 0-10 in a summative fashion. Higher summary score reflects more favorable state and lower summary score reflects the greatest room for improvement.
Change in Physical Activity questionnaire score | Baseline, 10-week, and 6 and 12 months after the program
  The brief Physical Activity "Vital Sign" (PAVS) will be used to determine if participants achieve the recommended amount of physical activity, with an additional question to assess use of yoga.Two questions are self-reported: 1) "How many days during the past week have you performed physical activity where your heart beats faster and your breathing is harder than normal for 30 minutes or more?" and 2) "How many days in a typical week do you perform activity such as this?" The responses are reported as days during the past week over days in a typical week, with scores ranging from 0 to 7 for each question. PAVS requires less than 30 seconds to administer and score
Change in Perceived Stress Scale score | Baseline, 10-week, and 6 and 12 months after the program
  The PSS-10 is a self-report instrument consisting of 10 items purported to assess "how unpredictable, uncontrollable, and overloaded respondents find their lives". Each of the items on the PSS-10 are rated on a 5-point Likert scale, ranging from 0 (never) to 4 (very often). The PSS-10 consisted of 6 positively (items 1, 2, 3, 6, 9 and 10: Positive factor) and 4 negatively (items 4, 5, 7 and 8: Negative factor) worded items. Negative worded items were re-coded during analysis. Total scores range from 0 to 40, with higher scores indicating higher levels of perceived stress
Change in Mindfulness and Mindful Eating Scale score | Baseline, 10-week, and 6 and 12 months after the program
  Mindful eating practices will be assessed using this Mindfulness and Mindful Eating tool. Domains of the 28-item questionnaire are: Disinhibition, Awareness, External Cues, Emotional Response, and Distraction. For all items, response options are "Never/Rarely," "Sometimes," "Often," and "Usually/Always". Each item is scored from 1 to 4, where higher scores signified more mindful eating. Each subscale score is calculated as the mean of items. The summary score is the mean of the 5 subscales.

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Bergquist, MD, Principal Investigator — Emory University
Locations (1):
- Emory Clinic, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual de-identified participant data - as reported in characteristics and results - will be shared
Supporting Information: SAP
Time Frame: Data will be available after publication and up to 36 months after publication
Access Criteria: Individual de-identified participant data will be shared through individual request for analyses pertaining to purpose of their study with investigators with approved institutional review committee studies